CLINICAL TRIAL: NCT02832583
Title: Efficacy of the Use of Autologous Platelet Rich Plasma Combined to Hyaluronic Acid Obtained With regenKit BCT-HA Cellular Matrix for Skin in Aesthetic Medicine
Brief Title: Autologous Platelet Rich Plasma Combined to Hyaluronic Acid Obtained With Regen-Kit BCT-HA in Aesthetic Medicine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regen Lab SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-A00718-39
Record Dates: First submitted 2016-07-05; First posted 2016-07-14 (Estimated); Last update posted 2016-10-03 (Estimated); Status verified 2016-09

CONDITIONS: Skin Wrinkling
Keywords: PRP, hyaluronic acid, mesotherapy, skin wrinkle, skin rejuvenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mesotherapy of PRP-HA into the cheeks (Experimental): Three sessions of PRP-HA prepared with RegenKit BCT-HA Cellular Matrix into each cheek separated by 1 month interval.
  Interventions: Device: Regenkit BCT-HA Cellular Matrix

INTERVENTIONS:
Device: Regenkit BCT-HA Cellular Matrix — To assess the efficacy of PRP-HA on skin rejuvenation, thirty one patients with chronological aging including wrinkles, dull and dry skin with loss of elasticity and firmness. The patients received three PRP-AH injection sessions 4 weeks apart into the cheeks.

SUMMARY:
The aim of this prospective study is to assess the efficacy of autologous Platelet Rich Plasma combined with Hyaluronic Acid prepared with RegenKit-BCT HA Cellular Matrix on skin rejuvenation. Thirty-one patients were included and received three PRP-AH injection sessions 4 weeks apart into the cheeks. The outcomes were assessed at baseline, 1, 3 and 6 months after the last injection session. Safety was assessed by reported adverse event analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 40 years with chronological aging
* Completed informed consent form

Exclusion Criteria:

* Pregnancy or breastfeeding
* Patients younger than 40 years
* Use of product or treatment aimed to improve skin rejuvenation over the last six months before study start,
* patients with known hypersensitivity to HA,
* patients with eczema flare-up,
* patients with active skin disorder infection including herpes virus infection, active hepatitis or human infection virus infection.
* Dermatological diseases affecting the face
* Auto-immune disease such as Hashimoto, rheumatoid arthritis.
* Malignancy with or without metastatic disease
* Chemotherapy
* Anticoagulant therapy

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-12; Primary Completion 2015-12 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Evaluate the changes of facial apparent overall assessed by FACE-Q scale. | 6 months
  Evaluate changes in facial apparent assessed by FACE-Q scale after 6 month of Autologous Platelet Rich Plasma combined to hyaluronic acid compared to baseline (before treatment)

SECONDARY OUTCOMES:
Evaluate the changes of skin elasticity assessed by the Cutometer® | 6 months
  Evaluate changes in skin elasticity assessed by the Cutometer® after 6 months of Autologous Platelet Rich Plasma combined to hyaluronic acid compared to baseline (before treatment).

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Hersant B, SidAhmed-Mezi M, Niddam J, La Padula S, Noel W, Ezzedine K, Rodriguez AM, Meningaud JP. Efficacy of autologous platelet-rich plasma combined with hyaluronic acid on skin facial rejuvenation: A prospective study. J Am Acad Dermatol. 2017 Sep;77(3):584-586. doi: 10.1016/j.jaad.2017.05.022. No abstract available. PMID 28807118